CLINICAL TRIAL: NCT01408810
Title: Histological and Endoscopic Evaluation of Remission Induced by Infliximab in Moderately to Severely Active Ulcerative Colitis Patients
Brief Title: Evaluation of Histologic and Endoscopic Remission Induced by Infliximab in Moderate to Severe Ulcerative Colitis
Acronym: HERICA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Grupo de Estudo da Doença Inflamatória Intestinal (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P06120
Record Dates: First submitted 2011-07-20; First posted 2011-08-03 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Ulcerative Colitis
Keywords: infliximab; ulcerative colitis; histologic remission
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Infliximab (Experimental): Infliximab 5 mg/Kg, I.V. at weeks 0, 2, 6 and every 8 weeks thereafter. The treatment should follow infliximab's Summary of Product Characteristics.
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — 5 mg/Kg, I.V. at weeks 0, 2, 6 and every 8 weeks thereafter
  Other Names: Remicade

SUMMARY:
The aim of this study is to assess the relationship between microscopic Geboes index of inflammation and clinical course of ulcerative colitis in patients treated with infliximab. The investigators propose to test the hypothesis if infliximab is able to induce histological remission and then change the clinical course of ulcerative colitis.

DETAILED DESCRIPTION:
Correlations between histologic disease activity and other assessments of clinical disease activity are not well established despite a good correlation being found between endoscopy and histology, especially during active ulcerative colitis (1,2). Endoscopic healing induced by infliximab in Crohn's disease patients was associated with a significant reduction in surgeries and hospitalizations (3). Histological recovery in ulcerative colitis is often incomplete and some studies have shown that microscopic evidence of inflammation is common even in patients with clinically and quiescent colitis assessed by sigmoidoscopy (4,5). Although this fact has not yet been completely elucidated, it is suggested that some patients with residual microscopic acute inflammation may be more prone to relapse (2). The prognostic importance of microscopic inflammation is unknown. Given that the rectum is always involved in ulcerative colitis and inflammatory activity is diffuse and restricted to the mucosa, the collection of samples from the rectal and sigmoid mucosa are potentially useful tools for evaluating disease severity. In addition, there is a strong correlation between the levels of calprotectin and the degree of inflammation as assessed by endoscopic and histologic criteria (6). Therefore, the measurement of faecal calprotectin and lactoferrin may also provide as valuable non-invasive tools to assess disease activity and optimize the treatment in UC patients.

Histologically, active disease is defined by the presence of neutrophils in conjunction with epithelial cell damage. Analysis generally relies on the examination of H & E-stained sections. Two samples are suggested as more appropriated because it is well-known that treatment may induce variations in the expression of inflammation intensity. Several histological scores were proposed, however, Geboes index (7) has been validated and tested for reproducibility and has 5 domains: structural change, chronic inflammatory infiltrate, lamina propria neutrophils and eosinophils, neutrophils in epithelium, crypt destruction and erosion or ulceration. The Geboes index has a more elaborated grading of crypt lesions and surface epithelial damage than other proposed indexes. The aim of this study is to assess the relationship between microscopic Geboes index of inflammation and clinical course of ulcerative colitis in patients treated with infliximab. The investigators propose to test the hypothesis if infliximab is able to induce histological remission and then change the clinical course of ulcerative colitis

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all the following inclusion criteria to be considered eligible:

  1. Must be eligible to start infliximab treatment according to the Portuguese approved Summary of Product Characteristics (SPC-See supplement 15.3)*
  2. Patients must be older than 18 years of age up to 65 years of age at the time of informed consent, of both gender and any race.
  3. Patients with moderate to severe UC - Mayo Score (6-12); endoscopic subscore ≥2
  4. Regarding the previous treatment exposure:

     4.1 Patients must have responded inadequately to corticosteroids at least a dose of 40mg/day with or without 5-ASA or patients steroid-dependent* 4.2- Patients must have responded inadequately to azathioprine or 6-MP (treatment with thiopurines must be at least 3 months in duration) or be intolerant to these agents.
  5. Patients must be naïve to infliximab or other anti-TNF agents
  6. No history of latent or active TB prior to screening. No signs or symptoms suggestive of active TB upon medical history and/or physical examination.
  7. Patients must be capable of providing written informed consent prior to trial entry.
  8. Subjects must be willing and able to adhere to visit protocol schedule and procedures.

     * Patients must have responded inadequately to corticosteroids at least a dose of 40mg/day with or without 5-ASA or patients steroid-dependent with a Mayo Score (6-12), endoscopic subscore >2. Steroid-dependent is defined as: patients unable to reduce steroids below 10mg/day within 3 months of starting steroids and patients who have a relapse within 3 months of stopping steroids.

Exclusion Criteria:

* 1- Any "Contraindication" as specified in the Portuguese infliximab approved Summary of Product Characteristics (See Supplement 15.3) 2- Patients with severe anemia (haemoglobin<8.0 g/dL) 3- Any malignancy in the past 5 years, including lymphoproliferative disorders 4- Existence of not removed adenomatous polyps 5- History of opportunistic infections in the last 6 months 6- Subjects who have a known viral infection such as CMV, HIV, HBV or HCV 7- Patients with a history of demyelinating diseases 8- Pregnant or breastfeeding women 9- Topical treatment with 5-ASA and steroids 10-Patients with only rectal involvement

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2011-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
histological remission | histological remission were assessed at week 8
  To assess if infliximab is able to induce histological remission in patients with moderately to severely active ulcerative colitis who have had an inadequate response to conventional therapy, including corticosteroids and 6-MP/AZA or who are intolerant or have medical contraindications for such therapies using Geboes criteria at week 8
Clinical response | clinical response were assessed at week 8
  To assess the clinical response in the above patients assessed by Mayo Score at week 8

SECONDARY OUTCOMES:
Histologic Efficacy assessment | baseline, week 8, week 30 and week 52.
  To assess the impact of infliximab histologically, four biopsies will be collected from distinct areas (two from rectum and two from sigmoid) from each patient
Correlate histological remission with mucosal healing,faecal calprotectin and lactoferrin levels,number of colectomies,number of hospitalizations,Number of clinical relapses | up to week 52
  Correlate histological remission with:
  Mucosal healing Faecal calprotectin and lactoferrin levels Number of colectomies up to week 52 Number of hospitalizations up to week 52 Number of clinical relapses up to week 52

CONTACTS AND LOCATIONS:
Overall Officials: Susana Lopes, MD, Principal Investigator — Hospital de São João; Francisco Portela, MD, Principal Investigator — Hospitais da Universidade de Coimbra; Paula Lago, MD, Principal Investigator — General Hospital of Santo António; José Cotter, MD, Principal Investigator — Hospital Nossa Senhora da Oliveira - Guimarães; Paula Peixe, MD, Principal Investigator — Centro Hospitalar Lisboa Ocidental Hospital Egas Moniz
Locations (1):
- Hospital de São João, Porto, Porto District, Portugal